CLINICAL TRIAL: NCT03714230
Title: The Trajectory of Functional Status During the First Year After ICU Admission.
Brief Title: Longitudinal Prospective Study in a Mixed ICU Population
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of California, San Francisco (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Professor, Oslo University Hospital
Other Study IDs: 2017/990
Record Dates: First submitted 2018-09-26; First posted 2018-10-22 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-04

CONDITIONS: Intensive Care Patients
Keywords: Functional status, Symptoms, Cognitive functioning, QOL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Longitudinal prospective observational multicenter study in a mixed population of intensive care unit (ICU) patients (n=650). The overall purpose of this research proposal is to increase the knowledge in how pre-morbid condition, symptoms during treatment, and selected clinical variables affect self-reported functional status during first year after an ICU admission.

DETAILED DESCRIPTION:
For this study data will be collected using self-report questionnaires for the long-term outcome (e.g functional status) and several covariates (e.g., cognition, anxiety and depression, PTSD, QOL, general symptoms, frailty). To retrieve baseline data from prior ICU admission, family members will be used as proxy reporters at inclusion. During treatment in the ICU, patients will be mapped for 5 pre-selected symptoms every day for 7 days, or until death or ICU discharge. Several clinical variables (e.g., SOFA score, pain score, level of sedation, mobilization, medication, mouth care) will be collected daily until maximum 7 days. Follow-up data will be collected at 3, 6 and 12 months after ICU admission using self-report questionnaires.

The predictive value of pre-morbid condition prior to ICU admission on functional status during the first year after an ICU admission will be investigated, when controlled for various clinical and demographic variables. As a secondary analyses, the present study will identify both the occurrence of symptoms as well as the severity and distress of each symptom, while in the ICU. Another secondary outcome that will be measured in this longitudinal study is the association between cognitive function one year after an ICU admission and various mental health variables (PTSD, anxiety and depression).

ELIGIBILITY:
Inclusion Criteria

* Patients that are > 18 years and
* Meet the criteria of Norwegian Intensive Register (NIR) for being an intensive care patient. The criteria include any on the following criteria:
* The need of mechanical ventilation, or
* The need of continuous inotropi, or
* 24 hours or more on an ICU, when continuous monitoring is needed, or
* Dies at the ICU within the first 24 hours, or
* Transferred to another ICU within the first 24 hours

Exclusion Criteria:

* Re-admissions to the ICU (within 72 hours from last ICU discharge)
* Pre-defined cognitive deficit (e.g. dementia)
* Homeless
* Unable to read and Write Norwegian
* Not included in the study within the first 48 hours since admission to the ICU

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample population is adults patients admitted to the ICU.
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
A cohort study on change of Functional Status during the first year after an ICU admission | September 2018- May 2020
  Data on functional status will be collected using PROMS (e.g Katz index and Lawton IADL) at baseline, and then after 3, 6 and 12 months.

SECONDARY OUTCOMES:
The investigation of 5 pre-selected symptoms during the ICU stay | September 2018 - December 2020
  A modified version of the Patient Symptom Survey (PSS) checklist will be used as self-report by the ICU patient when possible or by the clinical nurse as a proxy reporter.
Cognitive functioning one year after ICU admission in a mixed ICU population | September 2018 - December 2020
  Cognitive functioning will be measured using self-report with the Cognitive Failure Questionnaire, and proxy reported by IQCODE and CFQ at baseline.
Posttraumatic Stress Symptoms one year after ICU admission in a mixed ICU population, and the importance of hope | January 2020 - December 2021
  Posttraumatic stress symptoms will be measured using self-report with the Impact of event scale-revised questionnaire. Hope will be measured with the Herth Hope Index.

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, Professor, Principal Investigator — Oslo University Hospital and Oslo University
Locations (1):
- Oslo Univesity hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saltnes-Lillegard C, Rustoen T, Beitland S, Puntillo K, Hagen M, Lerdal A, Hofso K. Self-reported symptoms experienced by intensive care unit patients: a prospective observational multicenter study. Intensive Care Med. 2023 Nov;49(11):1370-1382. doi: 10.1007/s00134-023-07219-0. Epub 2023 Oct 9. PMID 37812229